CLINICAL TRIAL: NCT02931981
Title: Serum Dickkopf-4 as a Biomarker for the Diagnosis and Treatment of Gastrointestinal Stromal Tumor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GIST-DKK4
Record Dates: First submitted 2016-10-11; First posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Gastrointestinal Stromal Tumor
Keywords: DKK4; Gastrointestinal Stromal Tumor; Biomarker
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Surgical Procedures, Operative; Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: surgery or biopsy — Do radical surgery or biopsy to obtain a pathological result

SUMMARY:
Our study aims to evaluate the role of Dickkopf-4 as biomarkers in the treatment of gastrointestinal stromal tumor.

DETAILED DESCRIPTION:
To identify whether Dickkopf-4 (DKK4) could be a potential biomarker for diagnosis and prognosis in patients with gastrointestinal stromal tumor (GIST). Serum was collected from 50 patients with GIST. Serological levels of DKK4 were examined by enzyme-linked immunosorbent assay (ELISA). The sensitivity and specificity was compared with modified NIH risk criteria. A 3-year follow-up was monitored to evaluate the correlation between DKK4 serum levels and relapse-free or overall survival. The expression of DKK4 in GIST tumor tissues was also evaluated using immunohistochemistry staining.

ELIGIBILITY:
Inclusion Criteria:

* Primary gastrointestinal stromal tumor confirmed pathologically by surgery or biopsy
* Age from 18 - 70 years
* No serious organic and mental illness;

Exclusion Criteria:

* Pregnancy
* No pathologic result
* Suffering other malignancies at the same time.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gastrointestinal stromal tumor.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-10; Primary Completion 2016-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 3 years

SECONDARY OUTCOMES:
Relapse-free Survival | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics Committee of Renji Hospital, School of Medicine,Shanghai Jiaotong University, Shanghai, China